CLINICAL TRIAL: NCT05218798
Title: Comparison of the Different Tests Used to Measure Maximal Aerobic Capacity Among Slovenian Armed Forces
Brief Title: Enhancement of Physical and Combat Preparedness of SAF Members - Validation Study
Acronym: EPCPSAF-2021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Collaborators: Science and Research Centre Koper (Other)
Responsible Party: Principal Investigator, Armin Paravlic, Faculty of Sport, University of Ljubljana
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: EPCPSAF-2021-22-validation
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Physical Fitness; Cardio Respiratory Fitness; Aerobic Capacity; Physical Examination; Combat Preparedness

STUDY DESIGN:
Intervention Model Description: Crossover randomized validation study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects will be blinded for group allocation during testing procedures, including coaches (care provider), soldiers (participants) investigators, and outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Continous Treadmill Running Test (Active Comparator): One of the four testing conditions the subject will be allocated to is a Continous Treadmill Running Test. Vo2max will be measured by using A K4 b2 a portable gas analyzer (COSMED, Italy). The device provides reliable values for oxygen uptake (VO2), carbon dioxide production (VCO2), and pulmonary ventilation (VE) breath by breath. In addition, blood samples (20 μL) were collected from the earlobe for both tests (before, immediately after, 3 min after, and 5 min after the test) and the samples will be analyzed for blood lactate concentration ([LA-]).
  Interventions: Diagnostic Test: Cardio Respiratory Fitness testing
- Continous 2-mile run test (Active Comparator): One of the four testing conditions the subject will be allocated to is a Continous 2-mile run test. Vo2max will be measured by using A K4 b2 a portable gas analyzer (COSMED, Italy). The device provides reliable values for oxygen uptake (VO2), carbon dioxide production (VCO2), and pulmonary ventilation (VE) breath by breath. In addition, blood samples (20 μL) were collected from the earlobe for both tests (before, immediately after, 3 min after, and 5 min after the test) and the samples will be analyzed for blood lactate concentration ([LA-]).
  Interventions: Diagnostic Test: Cardio Respiratory Fitness testing
- 30-15 Intermittent Fitness Test - first trial (Active Comparator): Aerobic capacity will be measured using the field-based 30-15IFT test. This intermittent, incremental test consists of 30-second shuttle runs interspersed with 15-second active recovery periods. Running speed will be set at 8 km/h for the first 30-second run and increased by 0.5 km/h in each 30-second phase thereafter. The speed of the last successfully completed stage will be recorded as the test result, i.e. the maximum running speed (V) during IFT. Vo2max will be estimated by the following equation:
  Vo2max IFT (ml/min/kg) = 28.3 - 2.15G - 0.741A - 0.0357BM + 0.058A X VIFT + 1.03VIFT where G stands for subjects gender, A for age and BM for body mass, respectively.
  Interventions: Diagnostic Test: Cardio Respiratory Fitness testing
- 30-15 Intermittent Fitness Test - second trial (Active Comparator): The procedures will be the same as previously described
  Interventions: Diagnostic Test: Cardio Respiratory Fitness testing

INTERVENTIONS:
Diagnostic Test: Cardio Respiratory Fitness testing — In a randomized cross over designed study, we will measure Vo2max by using different tests:
  1. Continous Treadmill Running Test
  2. Continous 2-mile run test
  3. 30-15 Intermittent Fitness Test - first trial and second trial

SUMMARY:
The aim of the proposed project is to investigate the reliability, validity, and usefulness of the 30-15 intermittent fitness test in the Slovenian Armed Forces. We will compare the results obtained from a continuous treadmill running test, 2-mile run test, and 30-15IFT.

DETAILED DESCRIPTION:
Since the ability to perform military tasks depends on the physical fitness of soldiers (PF), one of the most commonly measured PF components during routine physical examinations is cardiorespiratory fitness (CRF). There are several tests used to measure CRF in the armed forces. Because of its simplicity, the most commonly used test of CRF is the 2-mile run test, but it has its own limitations when it comes to specificity of battlefield requirements, training prescription and optimization, and estimation of Vo2max. In combat situations, soldiers rarely run long distances on the battlefield. Therefore, the 2-mile run test does not appear to represent any specificity of combat. Furthermore, based on the data collected from this test, it is difficult to prescribe and optimize a training program for an individual subject. Therefore, the goal of the proposed project is to investigate the reliability, validity, and usefulness of the 30-15 intermittent fitness test in the Slovenian Armed Forces.

ELIGIBILITY:
Inclusion Criteria:

Members of Slovenian Armed Forces with no acute and/or chronic neuromuscular and skeletal injuries and/or any other chronic disease or conditions.

Exclusion Criteria:

older than 45 years of age acute and/or chronic neuromuscular and skeletal injuries the existence of any chronic disease or condition

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Maxima Oxygen Consumption (Vo2max) | 30 minutes
  Measure of maximal aerobic capacity (Vo2max)

SECONDARY OUTCOMES:
Maximal Running Speed | 30 minutes
  Maximal running speed achieved during different Vo2max testing batteries. The speed of the last successfully completed stage will be recorded as the test result, i.e. the maximum running speed (V) during IFT, or the last running speed reached during a continuous test will be defined as VTR
Tensiomyography (TMG) | 10 minutes
  We will use TMG to assess muscle fatigue from pre to post-different Vo2max testing procedures. The contractile properties of the individual muscles will be assessed by the non-invasive TMG method. We will measure knee extensor and flexors muscles of the dominant leg only.
Jumping ability | 10 minutes
  Countermovement and squat jumps will be used to assess muscle fatigue from pre to post-different Vo2max testing procedures. Jumping ability will be assessed by vertical jump tests, using a bilateral force plate (model 9260AA6, Kistler, Switzerland) with Kistler MARS software to record ground reaction force data.
D2 test | 5 minutes
  The D2 Test of Attention is a neuropsychological measure of selective and sustained attention and visual scanning speed. It is a paper and pencil test that asks participants to cross out any letter "d" with two marks around above it or below it in any order.
Stroop test | 2 minutes
  The stroop is a neuro-psychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute.

CONTACTS AND LOCATIONS:
Overall Officials: Janez Vodicar, Study Director — Faculty of Sport; Armin Paravlic, Principal Investigator — Faculty of Sport and Science and Research Centre Koper
Locations (1):
- Faculty of Sport, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
There is no plan for such an action. However, if the principal investigator and the project sponsor allow this aiming to collaborate on other projects, we will be interested to do so.

REFERENCES:
- [Result] Paravlic AH, Simunic B, Pisot R, Rauter S, Stuhec S, Vodicar J. The reliability, validity and usefulness of the 30-15 intermittent fitness test for cardiorespiratory fitness assessment in military personnel. Sci Rep. 2022 Sep 27;12(1):16087. doi: 10.1038/s41598-022-20315-3. PMID 36167789
- [Derived] Paravlic AH, Simunic B, Pisot R, Rauter S, Vodicar J. Reliability and validity of 30-15 intermittent fitness test for cardiorespiratory fitness assessment among infantry members of Slovenian armed forces: A study protocol. Front Psychol. 2022 Jul 22;13:894186. doi: 10.3389/fpsyg.2022.894186. eCollection 2022. PMID 35936328